CLINICAL TRIAL: NCT05837507
Title: Contribution of a Multimodal Digital Platform in the Management and Follow-up of Patients With Amyotrophic Lateral Sclerosis Treated With Non-invasive Ventilation: Randomized Controlled Study
Brief Title: Amyotrophic Lateral Sclerosis Non-invasive Ventilation Exchange
Acronym: ANEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Université Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL23_0054
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis (ALS); Non invasive ventilation; Telemonitoring; Telemedicine; Multidisciplinary approach
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, two-armed, interventional controlled study versus multicenter, open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): A group of 29 patients with ALS will be formed to the multimodal digital platform associated with Non Invasive Ventilation (NIV) and usual management
  Patients will be treated with NIV equipment from the manufacturer LOWENSTEIN and will benefit from the usual follow-up carried out at the reference center of Montpellier University Hospital.
  Interventions: Other: Telerehabilitation solution (m-Rehab); Other: Usual management including NIV.
- Control Comparator (Active Comparator): A group of 29 patients with ALS will be formed : control group following usual management including NIV.
  Patients will be treated with NIV equipment from the manufacturer LOWENSTEIN and will benefit from the usual follow-up carried out at the reference center of Montpellier University Hospital.
  Interventions: Other: Usual management including NIV.

INTERVENTIONS:
Other: Telerehabilitation solution (m-Rehab) — Patients in the experimental group will have access to a multimodal digital platform (m-Rehab®). The solution includes a website and an application available on smart phones for the patient and caregivers. Patients and caregivers will have access to educational content about the condition and its treatments, NIV compliance data, digital group educational workshops, secure messaging and video conferencing.
  All the professionals forming the patient's circle of care will be able to have access to the solution, after the patient's authorization. The circle of care, in a non-exhaustive way, includes specialist doctors, the general practitioner, the staff of the reference center of the Montpellier University Hospital, the physiotherapist, the speech therapist, the dietician and the psychologist.
  Arms: Experimental
Other: Usual management including NIV. — Usual management including NIV.

SUMMARY:
The median survival of patients with amyotrophic lateral sclerosis (ALS) is 3 to 5 years and mortality is mainly related to respiratory failure. Non-invasive ventilation (NIV) and multidisciplinary management improve the quality of life and survival of patients. However, patients have mobility difficulties related to the progressive worsening of functional disabilities. The research team hypothesize that the use of a multimodal digital platform, including in particular telemonitoring of NIV and teleconsultation, will slow down the evolution of the disabilities of patients with ALS and improve their quality of life.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a progressive neurodegenerative disease with a median life expectancy of 3 to 5 years. Respiratory failure due to alveolar hypoventilation is the main cause of mortality and respiratory impairment leads to a significant deterioration in quality of life.

Non-invasive ventilation (NIV) improves patient quality of life, improves gas exchange and improves patient survival. NIV should be initiated early, based on symptomatology and lung function, and monitored closely to adjust device parameters. NIV is a complex intervention that must be individualized for each patient.

In addition, multidisciplinary management involving different healthcare professionals, keeping the patient and caregivers at the center of the network, also allows for an improvement in the quality of life and survival of these patients.

However, patients with ALS have difficulty moving around and access to care becomes more complicated as the disease progresses. This phenomenon was increased during the COVID- 19 pandemic with a more rapid functional decline.

The development of new technologies should make it possible to rethink patient management, in particular through remote monitoring of NIV devices, teleconsultation, administration of questionnaires and better interprofessional organization. Several studies have confirmed the feasibility and acceptance of telemedicine solutions in this population.

In this project, The research team hypothesize that the use of a multimodal digital platform will slow the progression of disability in ALS patients and improve their quality of life, in particular by improving the quality of NIV and optimizing the coordination of a multidisciplinary team.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 30 and 85 years old
* Diagnosis of ALS
* Indication and acceptance of non-invasive ventilation
* Patient equipped with suitable equipment (tablet, computer, telephone, etc.) with an internet connection at home
* Patient able to read and understand the procedure, and able to express consent for the study protocol

Exclusion Criteria:

* Treatment with non-invasive ventilation in the previous three months
* Refusal/inability to use a smart phone or digital device
* Patient currently participating or having participated in the month preceding inclusion in another clinical interventional research that could impact the study, this impact is left to the discretion of the investigator.
* Subject under guardianship or curators
* Subject not affiliated to a social security scheme, or not a beneficiary of such a scheme.
* Subject deprived of liberty by judicial or administrative decision
* Pregnant, parturient, breastfeeding women
* Refusal to give consent

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Difference in change in functional abilities between the experimental and control groups over 6 months of follow-up. | Between baseline and 6 months
  Difference in variation of the functional capabilities assessed by the Amyotrophic lateral sclerosis functional rating scale (ALSFRS) score at Baseline (D0) and 6 months between the experimental group and the control group.
  A scale to determine different aspects of functionality in patients with ALS, minimum 0 points, maximum 48 points, derived from a questionnaire with 12 questions, each of which can yield up to 4 points, higher score indicates better functionality

SECONDARY OUTCOMES:
Difference in change in functional abilities between the experimental and control groups during 3 months of follow-up (Between 3 months and 6 months). | Between 3 months and 6 months
  Difference in variation of the functional capabilities assessed by the Amyotrophic lateral sclerosis functional rating scale (ALSFRS) score at 3 month and 6 month between the experimental group and the control group.
  A scale to determine different aspects of functionality in patients with ALS, minimum 0 points, maximum 48 points, derived from a questionnaire with 12 questions, each of which can yield up to 4 points, higher score indicates better functionality
Difference in change in functional abilities between the experimental and control groups during 3 months of follow-up (Between Baseline and 3 months). | Between Baseline and 3 months
  Difference in variation of the functional capabilities assessed by the ALSFRS score at Baseline (D0) and 3 month between the experimental group and the control group.
  A scale to determine different aspects of functionality in patients with ALS, minimum 0 points, maximum 48 points, derived from a questionnaire with 12 questions, each of which can yield up to 4 points, higher score indicates better functionality
Evolution of dyspnea between the 2 groups between baseline and 3 months | Between Baseline and 3 months
  Dyspnea assessed by modified Borg scale. Minimum is 0 (best). Maximum is 10 (worse).
Evolution of dyspnea between the 2 groups between baseline and 6 months | Between Baseline and 6 months
  Dyspnea assessed by modified Borg scale. Minimum is 0 (best). Maximum is 10 (worse).
Evolution of Quality of life between the 2 groups between baseline and 3 months | Between Baseline and 3 months
  Quality of life assessed by the EuroQol-5 Dimensions (EQ5D) scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Evolution of Quality of life between the 2 groups between baseline and 6 months | Between Baseline and 6 months
  Quality of life assessed by the EQ5D scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Evolution of evaluation of Anxiety and depression between the 2 groups between baseline and 3 months | Between Baseline and 3 months
  Anxiety and depression assessed by the Hospital Anxiety and Depression (HAD) scale.
  The HAD results in a score ranging from 0 (low anxiety or depression) to 21 (strong anxiety or depression).
Evolution of evaluation of Anxiety and depression between the 2 groups between baseline and 6 months | Between Baseline and 6 months
  Anxiety and depression assessed by the HAD scale. The HAD results in a score ranging from 0 (low anxiety or depression) to 21 (strong anxiety or depression).
Evolution of Patient satisfaction between the 2 groups between baseline and 3 months | Between Baseline and 3 months
  Patient satisfaction assessed by the CSQ-8 (Consumer satisfaction questionnaire) Minimal score is 8 and maximal score is 32. The best score is 32, that mean that patient is satisfied.
Evolution of Caregivers satisfaction between the 2 groups between baseline and 3 months | Between Baseline and 3 months
  Caregivers satisfaction assessed by the CSQ-8. Minimal score is 8 and maximal score is 32. The best score is 32, that mean that patient is satisfied.
Evolution of Patient satisfaction between the 2 groups between baseline and 6 months | Between Baseline and 6 months
  Patient satisfaction assessed by the CSQ-8. Minimal score is 8 and maximal score is 32. The best score is 32, that mean that patient is satisfied.
Evolution of Caregivers satisfaction between the 2 groups between baseline and 6 months | Between Baseline and 6 months
  Caregivers satisfaction assessed by the CSQ-8. Minimal score is 8 and maximal score is 32. The best score is 32, that mean that patient is satisfied.
Evolution of Anthropometric criteria between the 2 groups between baseline and 3 months (Weight measurements) | Between Baseline and 3 months
  Weight measurements
Evolution of Anthropometric criteria between the 2 groups between baseline and 3 months (BMI) | Between Baseline and 3 months
  BMI
Evolution of Anthropometric criteria between the 2 groups between baseline and 6 months (weight measurements) | Between Baseline and 6 months
  weight measurements
Evolution of Anthropometric criteria between the 2 groups between baseline and 6 months (BMI) | Between Baseline and 6 months
  BMI
Evaluation of the quality and tolerance of NIV between the 2 groups at 3 months | At 3 months
  The quality and tolerance of NIV assessed by the S3-NIV score. Score 0 to 10, lower units represent worse outcome.
Evaluation of the quality and tolerance of NIV between the 2 groups at 6 months | At 6 months
  The quality and tolerance of NIV assessed by the S3-NIV score. Score 0 to 10, lower units represent worse outcome.
Evaluation of the effectiveness of NIV between the 2 groups at 3 months assessed by nocturnal oximetry | At 3 months
  The effectiveness of NIV assessed by nocturnal oximetry
Evaluation of the effectiveness of NIV between the 2 groups at 6 months assessed by nocturnal oximetry | At 6 months
  The effectiveness of NIV assessed by nocturnal oximetry
Evaluation of the effectiveness of NIV between the 2 groups at 3 months assessed by nocturnal capnography | At 3 months
  The effectiveness of NIV assessed by nocturnal capnography
Evaluation of the effectiveness of NIV between the 2 groups at 6 months assessed by nocturnal capnography | At 6 months
  The effectiveness of NIV assessed by nocturnal capnography
Evaluation of the NIV parameters between the 2 groups at 3 months | At 3 months
  NIV parameters obtained using data from the machine report
Evaluation of the NIV parameters between the 2 groups at 6 months | At 6 months
  NIV parameters obtained using data from the machine report
Evaluation of survival between the 2 groups at 3 months | At 3 months
  Evaluation of survival between the 2 groups at 3 months
Evaluation of survival between the 2 groups at 6 months | At 6 months
  Evaluation of survival between the 2 groups at 6 months
Evaluation of time to first hospitalization between the 2 groups at 3 months | At 3 months
  recovery of hospitalization data
Evaluation of time to first hospitalization between the 2 groups at 6 months | At 6 months
  recovery of hospitalization data
Evaluation at 3 months in the experimental group of the Satisfaction of professionals with the digital solution | At 3 months
  Satisfaction of professionals with the digital solution by a VAS (Visual Analog Scale) of satisfaction
Evaluation at 6 months in the experimental group of the Satisfaction of professionals with the digital solution | At 6 months
  Satisfaction of professionals with the digital solution by a VAS (Visual Analog Scale) of satisfaction
Medico-economic evaluation: incremental cost-utility ratio | 6 months
  Utility will be derived from the EQ5D
Evaluation at 3 months in the experimental group of the Patient satisfaction with the digital solution | At 3 months
  Patient satisfaction with the digital solution assessed by a VAS (Visual Analog Scale) of satisfaction
Evaluation at 6 months in the experimental group of the Patient satisfaction with the digital solution | At 6 months
  Patient satisfaction with the digital solution assessed by a VAS (Visual Analog Scale) of satisfaction
Evaluation at 3 months in the experimental group of the caregiver satisfaction with the digital solution | At 3 months
  Caregiver satisfaction with the digital solution assessed by a VAS (Visual Analog Scale) of satisfaction
Evaluation at 6 months in the experimental group of the caregiver satisfaction with the digital solution | At 6 months
  Caregiver satisfaction with the digital solution assessed by a VAS (Visual Analog Scale) of satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Francois BUGHIN, MD, Study Director — University Hospital, Montpellier
Locations (2):
- France (2):
  - Uh Montpellier, Montpellier
  - Clinique du Millénaire, Montpellier

IPD SHARING:
Plan to Share IPD: Undecided